CLINICAL TRIAL: NCT00373659
Title: Prospective Optical Coherence Tomography (OCT) Imaging of Patients With Neovascular AMD Treated With Intra-Ocular Ranibizumab (Lucentis) (PrONTO) Study
Brief Title: An OCT-Guided Variable Dosing Regimen With Ranibizumab for the Treatment of Neovascular AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Philip J. Rosenfeld, MD, PhD, Professor of Ophthalmology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-FVF3102
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascularization; Age-related macular degeneration; Ranibizumab (Lucentis); Optical coherence tomography; Intravitreal injection
MeSH Terms: conditions — Neovascularization, Pathologic; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ranibizumab (Lucentis)

SUMMARY:
This study was designed to evaluate a variable dosing regimen with intravitreal ranibizumab for the treatment of patients with neovascular age-related macular degeneration (AMD) in the Prospective OCT Imaging of Patients with Neovascular AMD Treated with Intra-Ocular Ranibizumab (PrONTO) study.

DETAILED DESCRIPTION:
In this 2-year open-label, prospective, single-center, uncontrolled, investigator sponsored clinical study, neovascular AMD patients with subfoveal CNV (N=40) and a central retinal thickness of at least 300 µm as measured by optical coherence tomography (OCT) were enrolled to receive 3 consecutive monthly intravitreal injections of ranibizumab (0.5 mg). Thereafter, retreatment with ranibizumab was performed if one of the following changes were observed between visits: a loss of 5 letters in conjunction with fluid in the macula as detected by OCT, an increase in OCT central retinal thickness of at least 100 μm, new onset classic CNV, new macular hemorrhage, or persistent macular fluid following an injection of ranibizumab at the prior study visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Active primary or recurrent macular neovascularization secondary to age-related macular degeneration (AMD) involving the central fovea in the study eye with evidence of disease progression
* OCT central retinal thickness ≥ 300 microns
* Best corrected visual acuity, using ETDRS charts, of 20/40 to 20/400 (Snellen equivalent) in the study eye

Exclusion Criteria:

* More than 3 prior treatments with verteporfin photodynamic therapy
* Previous participation in a clinical trial (for either eye) involving antiangiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors)
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding day 0
* Subfoveal fibrosis or atrophy in the study eye
* History of vitrectomy surgery in the study eye
* Aphakia or absence of the posterior capsule in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity vs baseline
Change in OCT central retinal thickness vs baseline

SECONDARY OUTCOMES:
Number of injections over 1 year
Number of consecutive monthly injections until fluid-free
Injection free interval
Correlations of injection frequency with baseline lesion characteristics and visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Rosenfeld, MD PhD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Instiyute, Miami, Florida, United States